CLINICAL TRIAL: NCT05189405
Title: A 3 Year Retrospective Analysis of Fertility Clinic's of In Vitro Fertilization (IVF) in Comparison With INVOcell Intravaginal Culture (INVOcell IVC) Device
Brief Title: 3 Year Retrospective Analysis of IVF in Comparison With INVOcell
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: INVO Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-019
Record Dates: First submitted 2021-12-29; First posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- INVOcell IVC: IVF using intravaginal incubation with INVOcell device for embryo development.
  Interventions: Device: INVOcell IVC
- Traditional IVF (tIVF): Traditional IVF using laboratory equipment and incubators for embryo development

INTERVENTIONS:
Device: INVOcell IVC — Embryo development in intravaginal incubation
  Groups: INVOcell IVC

SUMMARY:
Retrospective chart review of data on the use of traditional IVF and INVOcell IVC collected from clinics using both technologies. The retrospective data will be utilized for a comparison of the two methods.

DETAILED DESCRIPTION:
The following aspects of data will be collected to support the analysis of the two methods

* Procedure details for including oil overlay and incubation time frame
* Characteristics of embryo quality and phase of development and transfer rates
* Clinical pregnancy rate
* Live birth rate Secondary: Data regarding safety
* Adverse events noted by the women that received IVF and INVOcell IVC
* Adverse events noted for the offspring

ELIGIBILITY:
Inclusion Criteria:

* Subjects that have received infertility treatment with either INVOcell IVC or standard IVF during the same timeframe. All subjects treated with the standard of care IVF method during the same timeframe that the center used INVOcell IVC were included in the retrospective data collection.

Exclusion Criteria:

* Not applicable

Ages: 18 Years to 42 Years | Sex: Female
Age Groups: Adult
Study Population: Subjects that have received infertility treatment with either INVOcell IVC or standard IVF during the same timeframe. All subjects treated with the standard of care IVF method during the same timeframe that the center used INVOcell IVC were included in the retrospective data collection.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2021-10-12 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Embryo development | 5 days
  Characteristics of embryo quality and phase of development and transfer rates
Clinical pregnancy rate | 5 days
  Clinical pregnancy rate
Live birth rate | 5 days
  Live birth rate

SECONDARY OUTCOMES:
Maternal Adverse Events | 5 days
  Adverse events noted by the women that received IVF and INVOcell IVC
Offspring adverse events | 5 days
  Adverse events noted for the offspring

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Carolina Conceptions, Raleigh, North Carolina
  - Piedmont Reproductive Endocrinology Group, Greenville, South Carolina
  - CARE Fertility, Bedford, Texas
  - THE NEW HOPE CENTER for Reproductive Medicine, Virginia Beach, Virginia